CLINICAL TRIAL: NCT04274491
Title: Predictors of Recovery Expectancy After Surgery for Pelvic Organ Prolapse
Brief Title: Predictors of Recovery Expectancy
Status: Completed | Type: Observational
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Andrew Doering, Co Principal Investigator, Indiana University
Other Study IDs: 2001849013
Record Dates: First submitted 2020-02-10; First posted 2020-02-18 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Pelvic Organ Prolapse; Surgery
Keywords: Recovery
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pelvic Organ Prolapse Surgery Patients: Participants with greater than or equal to stage II pelvic organ prolapse who are scheduled for reconstructive surgery will be recruited. Participants will be asked to complete a preoperative online survey regarding their health, recovery expectancy, and different roles. Additional online surveys will be send on postoperative days 14 and 42 to measure postdischarge surgical recovery

SUMMARY:
The purpose of this study is to identify factors that influence a person's expectations regarding recovery from pelvic organ prolapse surgery. This is important because a person's expectations regarding recovery from surgery help to predict how a person will actually recover. Our hypothesis is that women with multiple roles will have expectations of a longer surgical recovery time after surgery for pelvic organ prolapse after controlling for known predictors of recovery expectancies. Participants will complete a preoperative online survey. Additional online surveys will be send on postoperative days 14 and 42 to measure postdischarge surgical recovery.

ELIGIBILITY:
Inclusion Criteria:

* Patients with greater than or equal to stage II pelvic organ prolapse who are scheduled for reconstructive surgery.
* English speaking.
* Over the age of 18.
* Use email as a form of communication.
* Have a reliable internet connection at home.
* Have a computer/smartphone/tablet at home.

Exclusion Criteria:

* Non English speaking patients
* Patients without active email.
* Patients without access to reliable internet connection.
* Patients without access to computer/smartphone/tablet.
* Patients with less than stage II prolapse.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Patients with greater than or equal to stage II pelvic organ prolapse who are scheduled for reconstructive surgery.
Sampling Method: Non-Probability Sample
Enrollment: 202 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Recovery Expectancy | Participant will complete preoperative survey at 1 day (once surgery is scheduled).
  Expectation that recovery from surgery will be greater than 6 weeks from 0 to 100 percent where 100% indicates complete recovery within 6 weeks

SECONDARY OUTCOMES:
Post Discharge Recovery | Questionnaire will be completed on post op day #14
  Postdischarge Surgical Recovery Scale 13 which is validated tool for measuring postoperative recovery
Post Discharge Recovery | Questionnaire will be completed on post op day #42
  Postdischarge Surgical Recovery Scale 13 which is validated tool for measuring postoperative recovery

CONTACTS AND LOCATIONS:
Overall Officials: Michael Heit, MD, Principal Investigator — Indiana University
Locations (1):
- Indiana University Urogynecology, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Doering A, Hale D, Hamner J, Heit M. Predictors of Recovery Expectancy in Preparation for Pelvic Reconstructive Surgery in Women With Pelvic Organ Prolapse: A Prospective Cohort Study. Urogynecology (Phila). 2023 Jul 1;29(7):607-616. doi: 10.1097/SPV.0000000000001327. Epub 2023 Jan 12. PMID 36701635